CLINICAL TRIAL: NCT05765123
Title: A Pilot, Validation Study to Assess Sequential MRI Scanning on a 0.5 Tesla Upright Scanner as a Method to Determine Gastric Emptying Rate
Brief Title: Gastric Emptying Validation Pilot Study (MRI Val)
Acronym: MRIVal
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Luca Marciani, Professor, University of Nottingham
Other Study IDs: 40-0822
Record Dates: First submitted 2023-02-16; First posted 2023-03-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Dysfunction
Keywords: gastric emptying; Magnetic resonance imaging; '13-C acetate' breath test
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy male and female participants
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — A drink containing 75g of glucose together with 150mg carbon-13 sodium acetate in 300ml water

SUMMARY:
The primary aim of this study is to assess (in healthy volunteers) the rate at which a glucose drink leaves the stomach by sequential magnetic resonance imaging (MRI) of the stomach contents using a 0.5 tesla upright MRI scanner, and comparing with the rate derived from a standard method which uses a stable isotope tracer and breath testing. The main question it aims to answer are:

* Do MRI derived images of stomach contents at low magnetic field (0.5 Tesla) have sufficient resolution to provide a reproducible assessment of gastric emptying
* What is the agreement and relationship between the rate of gastric emptying determined from the 2 methods Participants will be asked to attend the imaging centre on one occasion in the morning after fasting from midnight and to sit within an upright MRI scanner for a period of approximately 140 minutes. Images of their stomach will be taken before and for 2 hours after consuming a drink containing glucose and a small amount of sodium acetate which contains a heavier form of carbon. Before each image is taken, participants will be asked to exhale into a 500ml bag to collect a breath sample.

DETAILED DESCRIPTION:
The rate at which food empties from the stomach is a key assessment made in appetite and metabolic research, as well as studies investigating gastrointestinal function in health and disease. This assessment can be achieved by measuring the volume of the stomach contents at timepoints after eating using magnetic resonance imaging (MRI) and calculating the gastric emptying rate from the decrease in volume which occurs over time. However, these measures are traditionally made when the individual is lying supine within the bore of the MRI machine and this postural position may impact the rate that food empties from the stomach. A low-field 0.5 Tesla 'upright' MRI scanner could address the problem of measuring gastric emptying rate when supine. However, the resolution of the images obtained are poorer than those obtained at higher field strengths (e.g. at 3 Tesla). The primary aim of this study is to compare gastric emptying kinetics assessed by sequential MR imaging of the stomach with a standard method which uses a stable isotope tracer (13-Carbon labelled sodium acetate) and breath testing. Twelve healthy, non-obese volunteers (18 to 60 years old) will attend the imaging centre on one occasion in the morning after fasting from midnight and sit within an upright MRI scanner for a period of approximately 140 minutes. Images of their stomach will be taken before and every 5 minutes for 1 hour, and every 10 minutes for the following hour, after consuming a drink containing glucose and 150mg of sodium acetate which contains a heavier (non-radioactive) form of carbon (carbon-13). Before each image is taken, participants will exhale into a 500ml bag to enable a breath sample to be collected. Breath samples will subsequently be analysed for carbon-13 enrichment of expired carbon dioxide (CO2) using mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (health status will be confirmed at screening).
* Able to fully comprehend the informed consent process and give informed consent.
* BMI <30 kg/m2

Exclusion Criteria:

* Known contraindication to MRI scanning (for example, pacemaker/implanted defibrillator, aneurysm clips, implanted programmable device, intra-ocular metallic fragment, claustrophobia)
* Major psychiatric, cognitive or mood disorder.
* Any other significant chronic medical conditions, including diabetes (type 1 and 2), asthma and epilepsy.
* Any acute major illness or surgery within one year prior to participation.
* Glucose intolerance (as assessed by a finger-prick test at screening).
* Having taken part in a research study in the last 3 months involving invasive procedures, ionising radiation or an inconvenience allowance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female adults
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
MRI gastric emptying rate (T50) | assessment made over 120 minutes (timepoints from 0 minutes to 120 minutes after consuming test drink)
  Gastric emptying rate (ml/min) derived from the decrease in volume of gastric contents
13-Carbon labelled Sodium Acetate Breath test gastric emptying rate (T50) | assessment made over 120 minutes (timepoints from 0 minutes to 120 minutes after consuming test drink)
  Gastric emptying rate derived (ml/min) from the rate of appearance of carbon 13 labelled CO2 in the breath

SECONDARY OUTCOMES:
Volume of gastric contents | assessed at timepoints from 0 minutes to 120 minutes after consuming the test drink (timepoints 0,5,10,15,20,25,30,35,40,45,50,55,60,70,80,90,100,110,and 120 minutes)
  Volume of gastric contents determined from MRI images (ml)
Carbon 13-enrichment of breath CO2 | assessed at timepoints from 0 minutes to 120 minutes after consuming the test drink (timepoints 0,5,10,15,20,25,30,35,40,45,50,55,60,70,80,90,100,110,and 120 minutes)
  carbon 13 labelled CO2 content in the breath measured using mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marciani, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Sir Peter Mansfield Imaging Centre, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No
anonymised data only shared where specific consent for data use in further studies has been given by the participants